CLINICAL TRIAL: NCT06804408
Title: Unpacking the "Mind" and "Body" Pathways of the Antidepressant Effect of Qigong in Older Adults: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, TSANG Hector Wing-Hong, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 15104721-1
Record Dates: First submitted 2025-01-07; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Qigong
MeSH Terms: interventions — Qigong

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Qigong (Experimental): 12-week training of Baduanjin (or named Eight-Section Brocades), with two sessions per week. Each session lasts for 60 min.
  Interventions: Behavioral: Qigong
- Mindfulness-based Training (Active Comparator): 12-week training of mindfulness-based breathing, walking, and stretching practices, with two sessions per week. Each session lasts for 60 min.
  Interventions: Behavioral: Mindfulness-based training
- Low-to-moderate Intensity Physical Exercise (Active Comparator): 12-week training of stretching, flexibility exercise, and balance exercise, with two sessions per week. Each session lasts for 60 min.
  Interventions: Behavioral: Low-to-moderate intensity physical exercise
- Waitlist (No Intervention): No training while the other three group are receiving training. Participants of this group are allowed to have Qigong, Mindfulness-based Training, or Low-to-moderate Intensity Physical Exercise after they complete all the assessments.

INTERVENTIONS:
Behavioral: Qigong — 12-week training of Baduanjin (or named Eight-Section Brocades), with two sessions per week. Each session lasts for 60 min.
  Arms: Qigong
Behavioral: Mindfulness-based training — 12-week training of mindfulness-based breathing, walking, and stretching practices, with two sessions per week. Each session lasts for 60 min.
  Arms: Mindfulness-based Training
Behavioral: Low-to-moderate intensity physical exercise — 12-week training of stretching, flexibility exercise, and balance exercise, with two sessions per week. Each session lasts for 60 min.
  Arms: Low-to-moderate Intensity Physical Exercise

SUMMARY:
The goals of the study are to explore the neurobiological mechanisms and cognitive benefits of qigong in older adults. The main research questions are:

* Does 12-week qigong training lead to significant enhancement in serum adiponectin, serum BDNF and significant reduction in salivary cortisol?
* Does 12-week qigong training bring significant improvement in global cognitive function?

Participants are older adults aged 60 or above. They were randomly assigned to qigong training, mindfulness training, physical exercise training, or wait-list which all last for 12 weeks. Their changes before and after the 12-week period in depressive symptoms, neurobiological markers, and cognitive functions are assessed.

ELIGIBILITY:
Inclusion Criteria:

* 60 years or older;
* With mild or severer levels of depressive symptoms as indicated by the Geriatric Depression Scale (GDS-8) scores of 5 or above, or Depression Anxiety and Stress Scale-21 (DASS-21) depression subscale scores of 4 or above
* Self-identified as physically stable and without life-threatening diseases.

Exclusion Criteria:

* With a history of practicing or receiving training of any form of mind-body or regular exercises (including tai chi, yoga, and qigong, or regular physical activity > 3 times/week) during the month prior to study enrollment
* Having changed medications or the dose of medications prescribed for their health condition in the month prior to study enrollment
* With severe cognitive or language impairment as defined as a score of less than 21 on Montreal Cognitive Assessment (MoCA-5min)
* Undergoing electroconvulsive therapy, psychotherapy, or psychoeducation for a psychological or psychiatric condition
* Unable to demonstrate satisfactory standing balance.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | Baseline and post-intervention (12 weeks after baseline)
  The eight-item Patient Health Questionnaire
Global cognitive function | Baseline and post-intervention (12 weeks after baseline)
  Montreal Cognitive Assessment

SECONDARY OUTCOMES:
Serum adiponectin | Baseline and post-intervention (12 weeks after baseline)
  Collected and assayed through peripheral blood sample
Serum BDNF | Baseline and post-intervention (12 weeks after baseline)
  Collected and assayed through peripheral blood sample
Salivary cortisol | Baseline and post-intervention (12 weeks after baseline)
  Collected and assayed through saliva sample
Attention | Baseline and post-intervention (12 weeks after baseline)
  Attention Network Task; Only collected from participants of Qigong and Waitlist groups
Inhibitory control | Baseline and post-intervention (12 weeks after baseline)
  Attention Network Task; Only collected from participants of Qigong and Waitlist groups
Working memory | Baseline and post-intervention (12 weeks after baseline)
  N-back Task; Only collected from participants of Qigong and Waitlist groups
ERP N2 amplitude | Baseline and post-intervention (12 weeks after baseline)
  ERP data recorded during Attention Network Task and N-back Task; Only collected from participants of Qigong and Waitlist groups
ERP P3 amplitude | Baseline and post-intervention (12 weeks after baseline)
  ERP data recorded during Attention Network Task and N-back Task; Only collected from participants of Qigong and Waitlist groups

CONTACTS AND LOCATIONS:
Locations (1):
- Hong Kong Polytechnic University, Department of Rehabilitation Sciences, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No